CLINICAL TRIAL: NCT00043342
Title: A Phase I/II Study of Interferon Gamma-1b by Subcutaneous Injection for the Treatment of Patients With Cystic Fibrosis
Brief Title: Study of Interferon Gamma-1b by Injection for the Treatment of Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GICF-002
Record Dates: First submitted 2002-08-07; First posted 2002-08-12 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; pulmonary impairment
MeSH Terms: conditions — Cystic Fibrosis | interventions — interferon gamma-1b

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: interferon gamma-1b — 100 or 200 mcg, SQ, 3x per week

SUMMARY:
The purpose of this research study is to evaluate the safety, tolerability, and efficacy of Interferon gamma-1b (IFN-gamma 1b) when administered by subcutaneous injection over a period of 4 weeks to patients with mild-to-moderate cystic fibrosis. Additionally, preliminary assessments on the effects of IFN-gamma 1b on lung function and other indicators of health will be made.

ELIGIBILITY:
* At least 6 years of age
* Diagnosis of cystic fibrosis (against certain criteria)
* Able to perform pulmonary (lung) function tests and participate in induced sputum procedures
* Pulmonary function values must meet certain minimal requirements
* Must have acceptable laboratory test results
* Cannot be on certain medications during and immediately prior to study
* Cannot have a history of unstable or deteriorating cardiac or neurologic disease

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2002-04; Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
change in sputum neutrophil count | 4 weeks

SECONDARY OUTCOMES:
change in predicted FEV1, sputum bacterial density, sputum levels of free neutrophil elastase, DNA and IL-8 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven Porter, MD, Study Director — InterMune